CLINICAL TRIAL: NCT03297476
Title: Early Precision Diagnosis and Relapse Prediction Technology Development in High-risk Acute Leukemia and Clinical Application
Brief Title: Clinical Application of Novel Panels for Early Precision Diagnosis and Relapse Prediction in High-risk Leukemia
Status: Completed | Type: Observational
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Ge Zheng, Director of Hematology Department, Zhongda Hospital
Other Study IDs: ZDYYGZ201708
Record Dates: First submitted 2017-08-15; First posted 2017-09-29 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Leukemia, Acute
MeSH Terms: conditions — Leukemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Patients' samples from bone marrow
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- high-risk group: Selected by "High-risk subtype detection panels"
  Interventions: Diagnostic Test: High-risk subtype detection panels
- non high-risk group: Selected by "High-risk subtype detection panels"
  Interventions: Diagnostic Test: High-risk subtype detection panels

INTERVENTIONS:
Diagnostic Test: High-risk subtype detection panels — The designed detection technology were used to identify the high-risk patients cohort.

SUMMARY:
Based on the investigator's previous data on risk classification for acute leukemia,the investigators will design a set of panels to detect the gene expression and genomic variants (SNPs, mutation, insertion, deletion and fusion genes, etc), and identify the high-risk subtypes of acute leukemia, such as Ph-like acute lymphoblastic leukemia. Furthermore, the target therapy (Tyrosine Kinase Inhibitors,et.al) will be used to treat the identified patients. In addition, more sensitive minimal residual disease (MRD) detection technology will be designed and used to detect the MRD in patients to early predict the disease relapse.

DETAILED DESCRIPTION:
patient eligibility criteria: newly diagnosed acute leukemia patients with clinical high-risk markers, reflactory and relapsed patients.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnostic acute lymphoblastic leukemia Be willing to start treatment

Exclusion Criteria:

* chronic leukemia

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with acute leukemia (newly diagnosis)
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
complete remission | From date of randomization or initial treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Patients achieve complete remission after initial treatment
relapse | From date of randomization or complete remission until the date of first documented relapse from any cause, whichever came first, assessed up to 100 weeks
  Patients' disease progress after complete remission

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Hematology, Zhongda Hospital Southeast University, Institute of Hematology Southeast University, Nanjing, Jiangsu, China